CLINICAL TRIAL: NCT04241939
Title: Brief Telephone Counseling and Numberless Scales to Overcome Weight Loss Barriers in Underserved Adolescents
Brief Title: Telephone Counseling and Numberless Scales to Overcome Barriers to Adolescent Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-0198; K12HD052023 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-01-27 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-01

CONDITIONS: Obesity
Keywords: Adolescent
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Numberless BDS and Modified-MI (Experimental): Use of numberless BDS (color coded), app, and motivational interviewing. Participants will weigh daily and receive weekly motivational interviewing at clinic visits and via a weekly phone call.
  Interventions: Behavioral: Numberless BDS; Behavioral: Modified Motivational Interviewing
- Digital Scale (Active Comparator): Use standard digital scale (number readout). Participants will weigh daily.
  Interventions: Behavioral: Digital Scale

INTERVENTIONS:
Behavioral: Numberless BDS — Participants perform daily weighing using a numberless BDS with feedback from app (color codes, challenges), in conjunction with modified motivational interviewing (clinic visits and weekly telephone calls), and the standard adolescent weight loss program.
  Arms: Numberless BDS and Modified-MI
Behavioral: Digital Scale — Participants perform daily weighing using a digital scale (number readout), in conjunction with standard adolescent weight loss program
  Arms: Digital Scale
Behavioral: Modified Motivational Interviewing — Modified motivational interviewing (clinic visits and weekly telephone calls), and the standard adolescent weight loss program.
  Arms: Numberless BDS and Modified-MI

SUMMARY:
This study tests the feasibility and acceptability of a numberless behavioral digital scale (BDS) intervention combined with motivational interviewing (MI) to affect lifestyle changes to promote weight loss in adolescents who are obese. Half of the participants will receive this intervention, while the other half will use a digital scale along with the standard adolescent weight loss program.

DETAILED DESCRIPTION:
The proposed pilot project seeks to enhance motivation for lifestyle change in adolescents who are obese. It will test a novel intervention that combines modified MI-based counseling and BDS. We will test the feasibility of the intervention over a 12-week period, with 24-week follow-up compared to use of standard digital scale. All participants will undergo the standard adolescent weight loss program, which includes monthly clinic visits with dietary and physical activity counseling. The MI intervention will include modified MI, brief weekly telephone reinforcement, and use of a BDS. The BDS with its mobile app offers daily feedback through colors, daily missions to promote healthy habits, and weekly healthy tips from nutritionists. In addition to the primary outcome of feasibility (daily weighing) investigators will also explore the intervention's effect on motivation, psychological outcomes and various aspects of feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 18 years
* BMI greater than or equal to 95th percentile for age and sex group or BMI greater than or equal to 35 kg/m^2
* Participant (not parent) is able to read and understand English (app is in English)
* Smartphone device with Wi-Fi and app capability
* Willingness to be randomized to any condition

Exclusion Criteria:

Age 19 years or older

* Developmental delay
* Inability to provide informed consent
* Any medical condition that, in the opinion of the PI, would place the participant at increased risk
* Use of an investigational agent in the 30 days prior to signing informed consent
* History of prior non-compliance or the presence or history of psychiatric condition (including drug or alcohol addiction) that would , in the opinion of the PI, make it difficult for the participant to comply with study procedures or follow instructions
* Females who are pregnant or lactating, by verbal report
* Pre-existing conditions (i.e paralysis, heart failure, severe autism or mental retardation, psychosis, etc.)
* Prisoners
* Lack of transportation

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Feasibility of Modified MI and BDS | 24 weeks
  Attendance at in-clinic visits, completion of weekly phone calls, and daily weighing based on BDS app data collected at 24 week assessment.
Acceptability of Modified MI and BDS | 24 weeks
  Number of participants in each group who are lost to follow-up

SECONDARY OUTCOMES:
Anthropometrics | 24 weeks
  Body Mass Index (BMI)
Bio-impedence measures | 24 weeks
  Measures body fat (%)
Anxiety | Change from 0 to 24 weeks
  Self-reported anxiety on a scale from 0 (not at all) to 3 (severely) using the Beck Anxiety Inventory
Depression | Change from 0 to 24 weeks
  Self-reported depression screening on a scale from 0 (not at all) to 3 (nearly every day) using the PHQ-9: Modified for Teens
Bio-impedence measures | 24 weeks
  Measures muscle mass (%)
Bio-impedence measures | 24 weeks
  Measures visceral fat (%)

CONTACTS AND LOCATIONS:
Overall Officials: Kanika Bowen-Jallow, MD, MMS, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - UTMB, League City, Texas
  - UTMB, Webster, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators will provide access to all data, regardless of publication, collected on this project. All external investigators must supply a written request identifying their research questions (s) and specifying the data they would like to analyze. The request must include a data security plan and explanation of how the data would be stored and who would have access.
Supporting Information: Study Protocol, SAP
Time Frame: Data available upon request
Access Criteria: All external investigators must supply a written request identifying their research questions (s) and specifying the data they would like to analyze. The request must include a data security plan and explanation of how the data would be stored and who would have access.